CLINICAL TRIAL: NCT02718508
Title: An e-Parenting Skills Intervention to Decrease Injured Adolescents' Alcohol Use
Acronym: e-Parenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael J. Mello, MD, MPH (Other)
Collaborators: Connecticut Children's Medical Center (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Michael J. Mello, MD, MPH, Director, Injury Prevention Center, Rhode Island Hospital
Organization: Rhode Island Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AA024185-01 (NIH)
Record Dates: First submitted 2016-03-02; First posted 2016-03-24 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Parenting; Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): All enrolled adolescents will continue to receive standard trauma center care, a brief intervention during their hospitalization by a trauma center social worker which is required by institutional policy.
- Standard Care plus e-Parenting Group (Experimental): The second group will continue to receive the same institutional standard care plus the parent will receive an e-parenting skills intervention consisting of: the online parent training program, Parenting Wisely (PW), plus text messaging and a web-based message board.
  Interventions: Behavioral: eParenting

INTERVENTIONS:
Behavioral: eParenting — The second group will continue to receive the same institutional standard care plus the parent will receive an e-parenting skills intervention consisting of: the online parent training program, Parenting Wisely (PW), plus text messaging and a web-based message board.
  Arms: Standard Care plus e-Parenting Group

SUMMARY:
The objective of this trial is to test feasibility and acceptability of an e-parenting skills intervention with parents of injured adolescent alcohol users (12-17 years old) as compared to standard care at three pediatric trauma centers. To examine these questions, the investigators will randomly assign adolescent and parent dyads (up to 75) to one of two groups. One group will continue to receive the institutional standard care of a brief alcohol intervention delivered by clinical staff to the adolescent with no parenting skills intervention. The second group will continue to receive the same institutional standard care plus the parent will receive an e-parenting skills intervention consisting of: the online parent training program, Parenting Wisely(PW), plus text messaging and a web-based message board. Study participants will be injured adolescents, 12-17 years old, admitted to the inpatient service of the trauma center, and with a positive CRAFFT (mnemonic acronym of first letters of key words in the screening tool) screen for alcohol use. Adolescents' alcohol use will be measured at study enrollment and at 3 and 6 months after discharge. Adolescents' alcohol related negative consequences will be measured at study enrollment for the 6 months prior to hospitalization and again at 6 months after hospital discharge. Parenting skills will also be assessed at 3 and 6 months.

DETAILED DESCRIPTION:
This study seeks to test the feasibility and acceptability of an e-parenting skills intervention at three pediatric trauma centers. The investigators will randomize up to 75 dyads of injured adolescents (12-17 years old) who screen positive for alcohol use and their parent to receive either standard trauma center care (a brief intervention with the adolescent) or standard trauma center care (a brief intervention with the adolescent) plus an e-parenting skills intervention consisting of a computerized intervention for parent skill building, a series of text messages and a web-based message board. The primary aim of this study is to determine the feasibility and acceptability of conducting the e-parenting intervention protocol across three pediatric trauma centers in preparation for a larger fully power trial. The central hypothesis for our future fully powered randomized control trial is that adolescents whose parents receive the e-parenting skills intervention will decrease their alcohol use and alcohol-related negative consequences over the 6 months following the intervention more than adolescents who receive only standard trauma center care. Therefore, a secondary aim of this proposal is to calculate a preliminary effect size that could be used, along with other relevant data, such as the acceptability data and findings in the literature, to calculate sample size in a future fully powered randomized control trial. The investigators will also examine adolescent's conjoint use of marijuana. This project advances translational research in collecting preliminary data on an e-parenting skills intervention that can be easily adopted with high fidelity across pediatric trauma centers. Its findings have the potential to directly impact best clinical practices for intervening with alcohol using injured adolescents

ELIGIBILITY:
Inclusion Criteria:

* adolescents, age 12-17, admitted to the trauma service
* medically stable
* a positive CRAFFT screen or lab screen for alcohol use or drug use
* ability to assent to study and have one parent consent
* adolescent and parent are English speaking

Exclusion Criteria:

* the adolescent is cognitively or emotionally unable to participate as determined by a trauma clinician
* the adolescent is suspected by the clinical staff of being a victim of child abuse (and referred to child protective services)
* the adolescent is being evaluated following a suicide attempt
* prior to admission, the adolescent is being treated for an alcohol or drug dependency
* adolescent is currently incarcerated

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability of an e-Parenting Skills Intervention | Up to 3 months
  Feasibility will be measured by parent data (number of Parenting Wisely logins and activities completed). Acceptability will be measured by the Systems Usability Scale (SUS) which rates parent ease of use of the program and the Consumer Satisfaction Questionnaire (CSQ) which rates level of parent satisfaction with treatment delivery and ability to manage child's behavior.

SECONDARY OUTCOMES:
Effects on Alcohol Use as assessed by Adolescent Drug Questionnaire (ADQ). | Up to 6 months
  Alcohol use will be measured by Adolescent Drug Questionnaire (number of drinking days and heavy drinking days in the past 3 months) among teen participants.
Effects on Drug use as assessed by Drug Use Questionnaire (DUQ). | Up to 6 months
  Drug use will be measured by Drug Use Questionnaire (number of days in the past 3 months teen participants used nicotine, marijuana, cocaine and other drugs).
Effects on Alcohol and Drug Related Problems as assessed by Add Health measures. | Up to 6 months
  Alcohol and drug related problems will be measured by the 9 questions from the Add Health survey (frequency of psychosocial and health consequences associated with alcohol and drug use over the prior 3 month period).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mello, MD, MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No